CLINICAL TRIAL: NCT06448754
Title: A Phase II, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Antitumor Activity of Volrustomig Priming Regimens in Combination With Other Anticancer Agents in Participants With Solid Tumors (eVOLVE-01)
Brief Title: Volrustomig Priming Regimens Exploratory Phase II Platform Study
Acronym: eVOLVE-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D798KC00001; 2023-509482-20-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-06-04; First posted 2024-06-07 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Solid Tumor; Programmed cell death-ligand-1; Tumor proportion score
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed; Ramucirumab; Paclitaxel

STUDY DESIGN:
Intervention Model Description: This platform study includes 2 substudies:
  Substudy 1 is randomized and Substudy 2 is non-randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Substudy 1: Arm 1A: Volrustomig dose regimen 1 + Carboplatin and Pemetrexed (Experimental): Volrustomig priming dose followed by volrustomig dosing regimen 1 in combination with carboplatin and pemetrexed.
  Interventions: Drug: Volrustomig; Drug: Carboplatin; Drug: Pemetrexed
- Substudy 1: Arm 1B: Volrustomig dose regimen 2 + Carboplatin and Pemetrexed (Experimental): Volrustomig priming dose followed by volrustomig dosing regimen 2 in combination with carboplatin and pemetrexed.
  Interventions: Drug: Volrustomig; Drug: Carboplatin; Drug: Pemetrexed
- Substudy 2: Arm 2A: Volrustomig dose regimen 2 +Ramucirumab + Carboplatin + Pemetrexed or Paclitaxel (Experimental): Volrustomig priming dose followed by volrustomig dosing regimen 2 in combination with ramucirumab and histology-specific chemotherapy (carboplatin+ either pemetrexed or paclitaxel).
  Interventions: Drug: Volrustomig; Drug: Carboplatin; Drug: Pemetrexed; Drug: Ramucirumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Volrustomig — Participants will receive volrustomig via intravenous (IV) infusion.
  Other Names: MEDI5752
Drug: Carboplatin — Participants will receive carboplatin via IV infusion.
Drug: Pemetrexed — Participants will receive pemetrexed via IV infusion.
Drug: Ramucirumab — Participants will receive ramucirumab via IV infusion.
  Arms: Substudy 2: Arm 2A: Volrustomig dose regimen 2 +Ramucirumab + Carboplatin + Pemetrexed or Paclitaxel
Drug: Paclitaxel — Participants will receive paclitaxel via IV infusion.
  Arms: Substudy 2: Arm 2A: Volrustomig dose regimen 2 +Ramucirumab + Carboplatin + Pemetrexed or Paclitaxel

SUMMARY:
Purpose of this study is to assess the safety, tolerability, pharmacokinetics, immunogenicity, and antitumor activity of volrustomig in combination with other anticancer drugs in participants with specified solid tumors.

DETAILED DESCRIPTION:
This Phase II, platform, open-label, multicenter study will evaluate the efficacy, safety, and tolerability of volrustomig in combination with anticancer drugs in various solid tumor types.

This platform study currently includes 2 substudies:

Substudy 1: metastatic non-small cell lung cancer (mNSCLC) (non-squamous [NSQ]). Participants will be randomized in two treatment arms: Arm 1A and Arm 1B.

Substudy 2: mNSCLC (squamous [SQ] or NSQ). Participants will enroll to the Arm 2A only.

All arms will test a volrustomig dosing in combination with chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with no deterioration.
* Life expectancy greater than or equal to (>=) 12 weeks.
* Adequate organ and bone marrow function.
* Body weight greater than (>) 35 kilograms (kg) at screening and at randomization.
* Histologically or cytologically documented NSQ NSCLC in substudy 1 and SQ or NSQ mNSCLC in substudy 2.
* Absence of sensitizing epidermal growth factor receptor (EGFR) mutations.
* Absence of documented tumor genomic alteration results from tests conducted as part of standard local practice in any other actionable driver oncogenes for which there are locally approved targeted 1L therapies.
* At least one measurable lesion not previously irradiated that can be accurately measured at baseline as >= 10 millimeter (mm) in the longest diameter.

Key Exclusion Criteria:

* Spinal cord compression.
* History of primary active immunodeficiency.
* Active or prior documented autoimmune or inflammatory disorders.
* Mixed small-cell lung cancer and NSCLC histology or sarcomatoid variant.
* Brain metastases unless asymptomatic, stable, and not requiring steroids for at least 14 days prior to start of study intervention. A minimum of 2 weeks must have elapsed between the end of radiation therapy and study enrollment.
* Prior chemotherapy or any other systemic therapy for Stage IV NSCLC. Participants who have received prior platinum-containing adjuvant, neoadjuvant, or definitive chemoradiation for local disease are eligible, provided that progression has occurred greater (>) 12 months from end of last therapy.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From screening (Days -28 to Day -1) up to 2 year 10 months
  The safety and tolerability of volrustomig in combination with other anticancer drugs in participants with specified solid tumors will be assessed.
Confirmed Objective Response rate (ORR) | Up to 2 year 10 months
  ORR is defined as the percentage of participants who have a confirmed complete response (CR) or confirmed partial response (PR), as per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to 2 year 10 months
  DCR is defined as the percentage of participants who have a CR or PR or who have stable disease (SD) after the date of randomization or first dose.
Duration of Response (DOR) | Up to 2 year 10 months
  DOR is defined as the time from the date of first documented response until the date of documented progression or death due to any cause (in the absence of progression).
Progression Free Survival (PFS) | Up to 2 year 10 months
  PFS is defined as the time from randomization or first dose until radiological progression or death due to any cause (in the absence of progression).
Overall Survival (OS) | Up to 2 year 10 months
  OS is defined as the time from randomization or first dose until the date of death due to any cause.
Serum Concentration of Volrustomig | Up to 2 year 10 months
  The serum concentrations volrustomig alone and when used in combination with other anticancer agents in participants with pre-specified solid tumors will be assessed.
Trough concentration (Ctrough) | Up to 2 year 10 months
  The trough concentrations volrustomig alone and when used in combination with other anticancer agents in participants with pre-specified solid tumors will be assessed.
Maximum Observed Concentration (Cmax) | Up to 2 year 10 months
  The serum concentrations volrustomig alone and when used in combination with other anticancer agents in participants with pre-specified solid tumors will be assessed.
Area Under the Curve (AUC) | Up to 2 year 10 months
  The AUC concentrations of volrustomig alone and when used in combination with other anticancer agents in participants with pre-specified solid tumors will be assessed.
Number of Participants with Positive Antidrug Antibodies (ADAs) | Up to 2 year 10 months
  The incidence of ADAs against volrustomig or other anticancer agents in serum will be assessed.

CONTACTS AND LOCATIONS:
Locations (64):
- United States (7):
  - Research Site, Los Angeles, California
  - Research Site, Grand Junction, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Tacoma, Washington
- Research Site, Montreal, Quebec, Canada
- China (5):
  - Research Site, Beijing
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Yantai
  - Research Site, Zhengzhou
- France (5):
  - Research Site, Bois-Guillaume
  - Research Site, Caen
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Montpellier
- Georgia (2):
  - Research Site, Batumi
  - Research Site, Tbilisi
- Greece (4):
  - Research Site, Athens
  - Research Site, Elaiones
  - Research Site, Piraeus
  - Research Site, Thessaloniki
- Italy (9):
  - Research Site, Genoa
  - Research Site, Meldola
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Perugia
  - Research Site, Rozzano
  - Research Site, Udine
  - Research Site, Verona
- Malaysia (3):
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
  - Research Site, Perai
- Portugal (2):
  - Research Site, Lisbon
  - Research Site, Porto
- Romania (3):
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Floreşti
- Serbia (3):
  - Research Site, Belgrade
  - Research Site, Kamenitz
  - Research Site, Kragujevac
- South Korea (3):
  - Research Site, Seongnam
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (9):
  - Research Site, A Coruña
  - Research Site, Alcorcón
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Santander
  - Research Site, Santiago de Compostela
  - Research Site, Valencia
- Switzerland (5):
  - Research Site, Basel
  - Research Site, Geneva
  - Research Site, Lausanne
  - Research Site, Winterthur
  - Research Site, Zurich
- Taiwan (3):
  - Research Site, Changhua
  - Research Site, New Taipei City
  - Research Site, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-leveldata from AstraZeneca group of companies sponsored clinical trials via therequest portal Vivli.org. All requests will be evaluated as per the AZ disclosurecommitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure."Yes",indicates that AZ are accepting requests for IPD, but this does not mean allrequests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitment smade to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment athttps://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure researchenvironmentVivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/